CLINICAL TRIAL: NCT05993351
Title: Correlating Advanced MRI Techniques With Neuropsychological Analysis and Immunosensing Assays for Assessment of Sport-related Mild Traumatic Brain Injuries (mTBI)
Brief Title: Objective Concussion Assessment Using MRI and Metabolomics
Status: Recruiting | Type: Observational
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Michael Noseworthy PhD, Director of MRI Research, Imaging Research Centre, St. Joseph's Healthcare Hamilton
Other Study IDs: Concussion MRI & recovery
Record Dates: First submitted 2023-08-12; First posted 2023-08-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-11

CONDITIONS: Concussion, Brain
Keywords: functional magnetic resonance imaging; diffusion tensor imaging; symptom tracking; sport-related concussions
MeSH Terms: conditions — Brain Concussion | interventions — Magnetic Resonance Imaging; Urination; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and saliva samples will be collected during each study visit for all participants to perform the metabolomic analyses. These samples will be stored in a -80 degree Celcius freezer until the time of batch analysis, for which the samples will be consumed. Any remaining biospecimens not consumed in the analyses will be disposed of appropraitely.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Concussion: Individuals who have recently sustained a concussion within the past 2-weeks.
  Interventions: Diagnostic Test: Magnetic resonance imaging (MRI); Diagnostic Test: Urine and saliva samples; Behavioral: Questionnaires
- Healthy Control: Individuals who have limited to no concussion history, and have not recently sustained a concussion.
  Interventions: Diagnostic Test: Magnetic resonance imaging (MRI); Diagnostic Test: Urine and saliva samples; Behavioral: Questionnaires

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging (MRI) — All participants will have 3 MRI scanning sessions to track brain health over time following the same protocol each time. The MRI sessions will occur acutely (<2 weeks post-concussion), 3-months and 6-months post-concussion. A series of MRI scans will be acquired including T1, T2, T2-FLAIR, SWI, ASL, rsfMRI, and DTI scans to characterize structural, microstructural, functional and tissue perfusion changes within the brain over time.
Diagnostic Test: Urine and saliva samples — At each study visit all participants will be asked to provide small urine and saliva samples for a metabolomic analysis using a high throughput multi-segment injection-capillary electrophoresis-mass spectrometry technology. This will allow for rapid non-targeted analysis of polar/hydrophilic metabolites, as well as non-polar/ionic lipids with stringent quality control.
Behavioral: Questionnaires — The Post-Concussion Symptom Scale (PCSS) and the Depression Anxiety Stress Scale (DASS-42) will be used to assess the self-reported presence and severity of known concussion-related symptoms.

SUMMARY:
Mild traumatic brain injury (mTBI), also referred to as concussions, affect millions of people around the world and can cause harmful long term effects. Unfortunately, concussions can be hard to diagnose and many people have lasting post-concussion symptoms such as headaches, difficulty concentrating, and light sensitivity. Recent studies have shown that advanced magnetic resonance imaging (MRI) techniques can identify subtle brain changes caused by a concussion. This study aims to track concussions over time measuring MRI brain scans and post-concussion symptoms to gain a better understand how the brain is affected in comparison to symptoms.

DETAILED DESCRIPTION:
Mild traumatic brain injuries (mTBI) are a major health concern due to the risk of short and long-term complications. In order to understand the effects of an TBI (also referred to as a concussion), studies have examined the physiological and cognitive impact of concussions on the brains of youth and collegiate athletes. Based on athletic-exposure (AE), the most concussions in the National Collegiate Athletics Association (NCAA) occur in Men's wrestling, Men's and Women's ice hockey, Men's football, and Women's soccer (Zuckerman et al. 2015). It has been estimated that 300 000 sport-related concussions (SRC) occur annually in the United States among youth and collegiate athletes (Coronado et al. 2015; Gessel et al. 2007; Langlois et al. 2006; Thurman et al. 1998). However, a SRC estimate would likely be grossly underestimated due to underreporting and failure to seek medical treatment (Karlin 2011; Kaut et al. 2003; Kerr et al. 2016; McCrea et al. 2004; Roozenbeek et al. 2013). In reality, the number of annual SRC could be as high as 1.6 to 3.8 million occurrences (Langlois et al. 2006).

Brain injuries are classified as mild, moderate or severe based on patient reported symptoms, cognitive impairment and structural damage visualized using medical imaging (Bodin et al. 2012; DeCuypere and Kilmo 2012; DeMatteo et al. 2010; Roozenbeek et al. 2013). A major challenge facing mTBI diagnosis has been standardizing assessment, predicting prognosis, and clearing people to return to work or sport. In order to more accurately diagnose and treat patients, healthcare providers require a better understanding of how to brain is affected acutely, and the timeline for when it returns to a pre-concussion state. Recent technological innovations show promise to supplement the current behavioural and psychological assessments. Current concussion and mTBI diagnosis are often based on tests that assess a patient's sensory feedback, mental cognition, motor control, and post-concussion symptoms (Bodin et al. 2012; DeCuypere and Klimo 2012).

To supplement symptom tracking, magnetic resonance imaging (MRI) has been shown in research to be an invaluable concussion tool. The health of brain white matter can be predicted based on the relativistic shape of the myelin surrounding axons and the diffusivity of water along the length of the axons by using a MRI technique called diffusion tensor imaging (DTI)(Asken et al. 2018; Jonkman et al. 2015). In addition, the function of brain grey matter can be assessed using functional magnetic resonance imaging (fMRI) by measuring the paramagnetic differences between oxygenated and deoxygenated blood, based on the Blood-Oxygen Level Dependent (BOLD) signal (Horn et al. 2014; Liu et al. 2018; Ogawa et al. 1990). Activated brain regions have a greater BOLD signal due to magnetic field inhomogeneities caused by changes in blood volume, blood flow, and local metabolism (Ogawa et al. 1990). An fMRI can be used to analyze brain resting state activation patterns, a primary connective system is the Default Mode Network (DMN)(Mak et al. 2017). The DMN has been shown to have decreased activity following a mTBI (Bonnelle et al. 2011; Zhou et al. 2012).

A serious issue surrounding head injuries is the need for a method to diagnose athletes immediately following the injury. The growing interest in using metabolomics for the discovery of clinically relevant biomarkers associated with mild traumatic brain injury (mTBI) could be a solution. However, most studies to date have relied exclusively on blood specimens and/or targeted metabolite panels involving small cohorts of patients without adequate replication, and validation of aberrant metabolic changes in circulation to independent MRI-based brain imaging (Fiandaca et al. 2018; Orešič et al. 2016). We propose to include an analysis of fasting saliva and urine specimens from mTBI patients for comprehensive metabolite profiling using high throughput multi-segment injection-capillary electrophoresis-mass spectrometry technology (DiBattista et al. 2019; Yamamoto et al. 2019), which allows for rapid non-targeted analysis of polar/hydrophilic metabolites, as well as non-polar/ionic lipids with stringent quality control (Azab et al. 2019).

This study aims to track concussion recovery over 6-months using clinical standards of concussion symptoms and objective MRI and metabolomics metrics. Concussion participants will complete three study visits: acutely within 2-weeks of a concussion, 3-month follow-up and 6-month follow-up. Participants will be recruited from St. Joseph's Healthcare Hamilton and local athletic organizations. The study protocol will be identical for all three study visits. Participants will complete the Post-Concussion Symptom Scale (PCSS) and Depression Anxiety Stress Scale (DASS-42) to measure the presence and self-reported severity of common post-concussion symptoms. The MRI data will be used to measure brain function (resting state fMRI) and microstructural properties (diffusion tenor imaging), while the metabolomics will measure if metabolites have abnormal presence or concentration post-concussion based on urine and saliva samples. These quantitative methods will be compared to the subjective concussion symptom scores to identify if brain and physiological abnormalities persist past symptom resolution, and if certain brain regions are more frequently affected by concussion. It is hypothesized that across all three time points that brain function will have decreased BOLD signal fractal complexity and network connectivity (representative of concussion-related injuries), and white matter damage will be present based on the primary DTI metric of fractional anisotropy. It is also hypothesized that post-concussion symptoms will be self-reported as resolved or almost resolved by the 3-month follow-up study visit.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 9-50
* Recently sustained a concussion (within the last 2 weeks)

Exclusion Criteria:

* Aged 8 and younger or 51 and older
* Unable to provide consent (e.g., poor English language skills, etc.)
* History of liver or kidney disease
* MRI contraindications:

  * Pacemaker
  * Stent
  * Joint prothesis
  * Implanted devices
  * Claustrophobia
  * Pregnant
  * Permanent piercings
* Chronic/abusive use of alcohol and/or illicit drugs
* Previous stroke or moderate/severe traumatic brain injury, subarachnoid hemorrhage, or intracranial hemorrhage
* Healthy control participants must not have a concussion history or recently sustained a concussion

Ages: 9 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants for this prospective observational cohort will include 50 individuals who have recently sustained a concussion within the last 2 weeks. Participants will primarily be recruited based on their involvement in collision or contact sport, causing sport-related concussions. Fifty healthy control participants will be recruited with the intention to have age, sex and athletic status matching to the concussion participants.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Functional brain characteristics | 45-minute MRI sessions acutely, 3-months and 6-months post-concussion
  Brain function will be examined based on the network connectivity and fractal complexity of the rsfMRI BOLD signal. This will be measured across known brain networks (e.g., Default Mode Network) and specific regions-of-interest (e.g., insula).
Microstructural brain characteristics | 45-minute MRI sessions acutely, 3-months and 6-months post-concussion
  Microstructural brain changes will be examined based on diffusion tensor imaging (DTI) metrics of fractional anisotropy, mean diffusivity, axial diffusivity, and radial diffusivity. This will be measured within specific regions-of-interest (e.g., insula).
Post-concussion symptoms | Acutely, 3-months and 6-months post-concussion
  Tracking of self-reported post-concussion symptoms using PCSS and DASS-42 questionnaires

SECONDARY OUTCOMES:
Metabolomics | Acutely, 3-months and 6-months post-concussion
  High throughput multi-segment injection-capillary electrophoresis-mass spectrometry technology will be used to analyze the urine and saliva samples to identify if any polar or non-polar metabolites are abnormal post-concussion, and that may indicate physiological markers for future assessment and treatment options.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Noseworthy, PhD, PEng, Principal Investigator — McMaster University; Dinesh A Kumbhare, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Imaging Research Center at St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Study data may be shared upon request to the research team.

REFERENCES:
- [Background] Asken BM, DeKosky ST, Clugston JR, Jaffee MS, Bauer RM. Diffusion tensor imaging (DTI) findings in adult civilian, military, and sport-related mild traumatic brain injury (mTBI): a systematic critical review. Brain Imaging Behav. 2018 Apr;12(2):585-612. doi: 10.1007/s11682-017-9708-9. PMID 28337734
- [Background] Azab S, Ly R, Britz-McKibbin P. Robust Method for High-Throughput Screening of Fatty Acids by Multisegment Injection-Nonaqueous Capillary Electrophoresis-Mass Spectrometry with Stringent Quality Control. Anal Chem. 2019 Feb 5;91(3):2329-2336. doi: 10.1021/acs.analchem.8b05054. Epub 2019 Jan 7. PMID 30570251
- [Background] Bodin, D., Yeates, K. O., & Klamar, K. (2012). Definition and Classification of Concussion. In J. N. Apps & K. D. Walter (Eds.), Pediatric and Adolescent Concussion (pp. 9-19). New York, NY: Springer New York. https://doi.org/10.1007/978-0-387-89545-1_2
- [Background] Bonnelle V, Leech R, Kinnunen KM, Ham TE, Beckmann CF, De Boissezon X, Greenwood RJ, Sharp DJ. Default mode network connectivity predicts sustained attention deficits after traumatic brain injury. J Neurosci. 2011 Sep 21;31(38):13442-51. doi: 10.1523/JNEUROSCI.1163-11.2011. PMID 21940437
- [Background] Coronado VG, Haileyesus T, Cheng TA, Bell JM, Haarbauer-Krupa J, Lionbarger MR, Flores-Herrera J, McGuire LC, Gilchrist J. Trends in Sports- and Recreation-Related Traumatic Brain Injuries Treated in US Emergency Departments: The National Electronic Injury Surveillance System-All Injury Program (NEISS-AIP) 2001-2012. J Head Trauma Rehabil. 2015 May-Jun;30(3):185-97. doi: 10.1097/HTR.0000000000000156. PMID 25955705
- [Background] Decuypere M, Klimo P Jr. Spectrum of traumatic brain injury from mild to severe. Surg Clin North Am. 2012 Aug;92(4):939-57, ix. doi: 10.1016/j.suc.2012.04.005. Epub 2012 Jun 5. PMID 22850156
- [Background] Dematteo CA, Hanna SE, Mahoney WJ, Hollenberg RD, Scott LA, Law MC, Newman A, Lin CY, Xu L. "My child doesn't have a brain injury, he only has a concussion". Pediatrics. 2010 Feb;125(2):327-34. doi: 10.1542/peds.2008-2720. Epub 2010 Jan 18. PMID 20083526
- [Background] DiBattista A, McIntosh N, Lamoureux M, Al-Dirbashi OY, Chakraborty P, Britz-McKibbin P. Metabolic Signatures of Cystic Fibrosis Identified in Dried Blood Spots For Newborn Screening Without Carrier Identification. J Proteome Res. 2019 Mar 1;18(3):841-854. doi: 10.1021/acs.jproteome.8b00351. Epub 2019 Jan 7. PMID 30507207
- [Background] Fiandaca MS, Mapstone M, Mahmoodi A, Gross T, Macciardi F, Cheema AK, Merchant-Borna K, Bazarian J, Federoff HJ. Plasma metabolomic biomarkers accurately classify acute mild traumatic brain injury from controls. PLoS One. 2018 Apr 20;13(4):e0195318. doi: 10.1371/journal.pone.0195318. eCollection 2018. PMID 29677216
- [Background] Gessel LM, Fields SK, Collins CL, Dick RW, Comstock RD. Concussions among United States high school and collegiate athletes. J Athl Train. 2007 Oct-Dec;42(4):495-503. PMID 18174937
- [Background] Horn A, Ostwald D, Reisert M, Blankenburg F. The structural-functional connectome and the default mode network of the human brain. Neuroimage. 2014 Nov 15;102 Pt 1:142-51. doi: 10.1016/j.neuroimage.2013.09.069. Epub 2013 Oct 4. PMID 24099851
- [Background] Jonkman LE, Rosenthal DM, Sormani MP, Miles L, Herbert J, Grossman RI, Inglese M. Gray Matter Correlates of Cognitive Performance Differ between Relapsing-Remitting and Primary-Progressive Multiple Sclerosis. PLoS One. 2015 Oct 20;10(10):e0129380. doi: 10.1371/journal.pone.0129380. eCollection 2015. PMID 26485710
- [Background] Karlin AM. Concussion in the pediatric and adolescent population: "different population, different concerns". PM R. 2011 Oct;3(10 Suppl 2):S369-79. doi: 10.1016/j.pmrj.2011.07.015. PMID 22035679
- [Background] Kaut KP, DePompei R, Kerr J, Congeni J. Reports of head injury and symptom knowledge among college athletes: implications for assessment and educational intervention. Clin J Sport Med. 2003 Jul;13(4):213-21. doi: 10.1097/00042752-200307000-00004. PMID 12855923
- [Background] Kerr ZY, Register-Mihalik JK, Kroshus E, Baugh CM, Marshall SW. Motivations Associated With Nondisclosure of Self-Reported Concussions in Former Collegiate Athletes. Am J Sports Med. 2016 Jan;44(1):220-5. doi: 10.1177/0363546515612082. Epub 2015 Nov 18. PMID 26582799
- [Background] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222
- [Background] Liu X, Zhang N, Chang C, Duyn JH. Co-activation patterns in resting-state fMRI signals. Neuroimage. 2018 Oct 15;180(Pt B):485-494. doi: 10.1016/j.neuroimage.2018.01.041. Epub 2018 Feb 21. PMID 29355767
- [Background] Mak LE, Minuzzi L, MacQueen G, Hall G, Kennedy SH, Milev R. The Default Mode Network in Healthy Individuals: A Systematic Review and Meta-Analysis. Brain Connect. 2017 Feb;7(1):25-33. doi: 10.1089/brain.2016.0438. Epub 2017 Jan 9. PMID 27917679
- [Background] McCrea M, Prichep L, Powell MR, Chabot R, Barr WB. Acute effects and recovery after sport-related concussion: a neurocognitive and quantitative brain electrical activity study. J Head Trauma Rehabil. 2010 Jul-Aug;25(4):283-92. doi: 10.1097/HTR.0b013e3181e67923. PMID 20611046
- [Background] Ogawa S, Lee TM, Nayak AS, Glynn P. Oxygenation-sensitive contrast in magnetic resonance image of rodent brain at high magnetic fields. Magn Reson Med. 1990 Apr;14(1):68-78. doi: 10.1002/mrm.1910140108. PMID 2161986
- [Background] Oresic M, Posti JP, Kamstrup-Nielsen MH, Takala RSK, Lingsma HF, Mattila I, Jantti S, Katila AJ, Carpenter KLH, Ala-Seppala H, Kyllonen A, Maanpaa HR, Tallus J, Coles JP, Heino I, Frantzen J, Hutchinson PJ, Menon DK, Tenovuo O, Hyotylainen T. Human Serum Metabolites Associate With Severity and Patient Outcomes in Traumatic Brain Injury. EBioMedicine. 2016 Oct;12:118-126. doi: 10.1016/j.ebiom.2016.07.015. Epub 2016 Jul 15. PMID 27665050
- [Background] Roozenbeek B, Maas AI, Menon DK. Changing patterns in the epidemiology of traumatic brain injury. Nat Rev Neurol. 2013 Apr;9(4):231-6. doi: 10.1038/nrneurol.2013.22. Epub 2013 Feb 26. PMID 23443846
- [Background] Thurman DJ, Branche CM, Sniezek JE. The epidemiology of sports-related traumatic brain injuries in the United States: recent developments. J Head Trauma Rehabil. 1998 Apr;13(2):1-8. doi: 10.1097/00001199-199804000-00003. PMID 9575252
- [Background] Yamamoto M, Pinto-Sanchez MI, Bercik P, Britz-McKibbin P. Metabolomics reveals elevated urinary excretion of collagen degradation and epithelial cell turnover products in irritable bowel syndrome patients. Metabolomics. 2019 May 20;15(6):82. doi: 10.1007/s11306-019-1543-0. PMID 31111238
- [Background] Zhou Y, Milham MP, Lui YW, Miles L, Reaume J, Sodickson DK, Grossman RI, Ge Y. Default-mode network disruption in mild traumatic brain injury. Radiology. 2012 Dec;265(3):882-92. doi: 10.1148/radiol.12120748. PMID 23175546
- [Background] Zuckerman SL, Kerr ZY, Yengo-Kahn A, Wasserman E, Covassin T, Solomon GS. Epidemiology of Sports-Related Concussion in NCAA Athletes From 2009-2010 to 2013-2014: Incidence, Recurrence, and Mechanisms. Am J Sports Med. 2015 Nov;43(11):2654-62. doi: 10.1177/0363546515599634. Epub 2015 Sep 1. PMID 26330572